CLINICAL TRIAL: NCT02807844
Title: A Phase Ib/II, Open Label, Multicenter Study of MCS110 in Combination With PDR001 in Patients With Advanced Malignancies
Brief Title: Phase Ib/II Study of MCS110 in Combination With PDR001 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMCS110Z2102; 2016-000210-29 (EudraCT Number)
Record Dates: First submitted 2016-06-17; First posted 2016-06-21 (Estimated); Results first posted 2021-08-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Triple Negative Breast Cancer; Pancreatic Carcinoma; Melanoma; Endometrial Carcinoma
Keywords: Triple negative breast cancer; Pancreatic carcinoma; Melanoma; Endometrial Carcinoma; Immuno oncology; Monoclonal antibody; PDR001; MCS110; Advanced malignancies; metasteses; advanced cancer; malignant
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Pancreatic Neoplasms; Melanoma; Endometrial Neoplasms | interventions — Macrophage Colony-Stimulating Factor; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W (Experimental): Phase Ib: MCS110 1 mg/kg every 3 weeks (Q3W) + PDR001 100 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W (Experimental): Phase Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W (Experimental): Phase Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W (Experimental): Phase Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W (Experimental): Phase Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W (Experimental): Phase Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
  Interventions: Drug: MCS110; Drug: PDR001
- Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC (Experimental): Phase II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - Triple negative breast cancer (TNBC)
  Interventions: Drug: MCS110; Drug: PDR001
- Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC (Experimental): Phase II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - Pancreatic cancer (PC)
  Interventions: Drug: MCS110; Drug: PDR001
- Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC (Experimental): Phase II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - Endometrial cancer (EC)
  Interventions: Drug: MCS110; Drug: PDR001
- Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME (Experimental): Phase II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - Melanoma (ME)
  Interventions: Drug: MCS110; Drug: PDR001

INTERVENTIONS:
Drug: MCS110 — MCS110 and PDR001 - for administration once every 3 weeks via i.v. infusion.
  Other Names: colony-stimulating factor-1 [CSF-1])
Drug: PDR001 — MCS110 and PDR001 - for administration once every 3 weeks via i.v. infusion.

SUMMARY:
The purpose of this study of MCS110 with PDR001 was to characterize the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and antitumor activity of the combination of MCS110 with PDR001 in adult patients with solid tumors.

DETAILED DESCRIPTION:
Combined treatment with MCS110 and PDR001 was expected to result in Tumor-associated macrophages (TAM) depletion, enhanced T-cell activation and synergistic antitumor activity in the clinical setting.

This study was a Phase Ib/II, multi-center, open label study starting with a Phase Ib dose escalation part followed by a Phase II part. MCS110 and PDR001 were administered i.v. Q3W until the patient experienced unacceptable toxicity, progressive disease as per irRC and/or treatment was discontinued at the discretion of the investigator or the patient. Patients were not to discontinue treatment based on progressive disease per Response evaluation criteria in solid tumors (RECIST) v1.1. During the Phase Ib part of the study, cohorts of patients were treated with increasing doses of MCS110 and PDR001 every 3 weeks until a Recommended Phase 2 Dose (RP2D) was determined for this treatment combination.

To assure that the combination RP2D did not exceed the Maximum tolerated dose (MTD), the combination MCS110 and PDR001 dose escalation was guided by a Bayesian logistic regression model (BLRM) with overdose control (EWOC) principle based on dose limiting toxicity data in the context of available safety, Pharmacokinetics (PK) and Pharmacodynamics (PD) information. Once the MTD and/or RP2D was declared, additional patients were enrolled in the Phase II part in order to assess the preliminary anti-tumor activity of MCS110 in combination with PDR001 in anti-PD1/PD-L1-naive triple negative breast cancer (TNBC), pancreatic (PC), endometrial carcinoma (EC) and anti PD1/PD-L1-resistance melanoma (ME).

ELIGIBILITY:
Main Inclusion Criteria:

* Signed informed consent prior to any procedures
* Phase Ib part: Adult patients with advanced melanoma, endometrial carcinoma, pancreatic or TNBC, with measurable or non-measurable disease who have progressed despite standard therapy or are intolerant of standard therapy, or for whom no standard therapy exists.
* Phase II part: Adult patients with advanced solid tumors who have received standard therapy (no more than 3 prior lines of treatment) or are intolerant of standard therapy, have progressed following their last prior therapy, and fit into one of the following groups:

  * Group 1: TNBC who did not receive prior anti-PD-1/PD-L1 treatment
  * Group 2: Pancreatic adenocarcinoma who did not receive prior anti-PD-1/PD-L1 treatment
  * Group 3: Endometrial carcinoma who did not receive prior anti-PD-1/PD-L1 treatment
  * Group 4: Melanoma who progressed on prior anti-PD-1/PD-L1 treatment.

Main Exclusion Criteria:

* Patients with the following:

  * Symptomatic central nervous system (CNS) metastases or those requiring local CNS-directed therapy.
  * Abnormal liver, renal, or blood lab values.
  * Impaired cardiac function or clinically significant cardiac disease.
  * Active autoimmune disease or documented autoimmune disease within 3 years of screening.
  * Active infection requiring antibiotic therapy.
  * Known HIV, active hepatitis B or C virus.
  * Concurrent malignant disease.
* Patients who received systemic anticancer therapy, major surgery, or radiotherapy within 2 weeks of study treatment, or live vaccines within 4 weeks of study treatment.
* Patients requiring chronic treatment with systemic steroid therapy or any immunosuppressive therapy.
* Patients who used hematopoietic colony-stimulating growth factors within 2 weeks of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-06-29 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (18):
- United States (4):
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - The West Clinic, Germantown, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, HUS, Finland
- Novartis Investigative Site, Saint-Herblain, France
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Hong Kong, Hong Kong
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Novartis Investigative Site, Seoul, South Korea
- Spain (2):
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Madrid
- Switzerland (3):
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Geneva
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Ahmed J, Stephen B, Yang Y, Kwiatkowski E, Ejezie CL, Pant S. Phase Ib/II Study of Lacnotuzumab in Combination with Spartalizumab in Patients with Advanced Malignancies. J Immunother Precis Oncol. 2024 May 2;7(2):73-81. doi: 10.36401/JIPO-23-16. eCollection 2024 May. PMID 38721402

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Started | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 2
Not completed — Death | 0 | 0 | 2 | 4 | 1 | 2 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — Progressive disease | 5 | 12 | 8 | 8 | 3 | 8 | 14 | 17 | 19 | 15
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME | Total
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20 | 141
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 9 | 8 | 10 | 5 | 8 | 20 | 11 | 9 | 12 | 95
  >=65 years | 3 | 3 | 4 | 3 | 1 | 3 | 0 | 9 | 12 | 8 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (14.72) | 56.9 (11.13) | 59.3 (9.94) | 55.4 (10.03) | 57.3 (14.02) | 58.6 (11.13) | 50.0 (8.29) | 61.5 (11.33) | 62.8 (10.13) | 60.7 (13.15) | 58.5 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 6 | 8 | 4 | 6 | 20 | 8 | 21 | 9 | 96
  Male | 2 | 2 | 6 | 5 | 2 | 5 | 0 | 12 | 0 | 11 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 2 | 1 | 2 | 5 | 4 | 4 | 7 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  White | 5 | 12 | 10 | 11 | 5 | 9 | 14 | 14 | 14 | 12 | 106
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Percentage of Participants With Adverse Events, as a Measure of Safety
Description: Phase Ib: To characterize the safety and tolerability of MCS110 in combination with PDR001 in patients with advanced solid malignancies and to identify a recommended dose combination for Phase II.
Time Frame: From start of treatment to a maximum timeframe of 116.4 weeks for phase Ib
Population: Safety Analysis Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Participants
  Adverse events (AEs) - all grades | 6 | 12 | 12 | 13 | 6 | 11
  Adverse events - Treatment-related - all grades | 6 | 12 | 11 | 8 | 6 | 8
  Serious Adverse Events (SAEs) - all grades | 3 | 4 | 4 | 7 | 2 | 5
  SAEs - Treatment-related - all grades | 0 | 1 | 0 | 0 | 2 | 1
  Fatal SAEs - all grades | 0 | 0 | 0 | 2 | 0 | 0
  Fatal SAEs - Treatment-related - all grades | 0 | 0 | 0 | 0 | 0 | 0
  AEs leading to discontinuation - all grades | 0 | 0 | 0 | 0 | 2 | 1
  AEs leading to discontinuation - Treatment-related - all grades | 0 | 0 | 0 | 0 | 2 | 1
  AEs leading to dose adjustment / interruption - all grades | 4 | 4 | 4 | 2 | 2 | 6
  AEs requiring additional therapy - all grades | 6 | 12 | 10 | 12 | 4 | 10

2. Primary Outcome: Phase II : Overall Response Rate (ORR) - Per RECIST v1.1
Description: Overall Response Rate (ORR) is defined as the proportion of patients with a best overall response assessed by CT scan or MRI of complete response (CR), disappearance of all measurable and non-measurable lesions or partial response (PR), at least a 30% decrease in the sum of diameter of all measurable lesions, taking as reference the baseline sum of diameters,. based on local Investigator assessment, as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1)
Time Frame: 4 years
Population: Full Analysis Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 5 [0.3 to 21.6] | 0 [0.0 to 13.9] | 9.5 [1.7 to 27.1] | 0 [0.0 to 13.9]

3. Primary Outcome: Phase II : Bayesian Inference of Overall Response Rate (ORR) - Per RECIST v1.1 - Mean
Description: Overall Response Rate (ORR) is defined as the proportion of patients with a best overall response assessed by CT scan or MRI of complete response (CR), disappearance of all measurable and non-measurable lesions or partial response (PR), at least a 30% decrease in the sum of diameter of all measurable lesions, taking as reference the baseline sum of diameters,. based on local Investigator assessment, as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) - mean (FAS)
Time Frame: 4 years
Population: Full Analysis Set. Since objective responses are rare in advanced pancreatic cancer and that long lasting stable disease is considered beneficial to patients, clinical benefit rate (confirmed objective response or SD>4 months) was used as the primary endpoint for antitumor activity in this study changed from objective response to for this patient population.
Measure: Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 6.7 [0.8 to 17.1] | NA [NA to NA] — Bayesian inference of Clinical Benefit Rate was measured for this arm instead - see Bayesian inference of Clinical Benefit Rate - per RECIST v1.1- mean results | 10.8 [2.6 to 23.1] | 0.8 [0 to 4.5]

4. Primary Outcome: Phase II: Clinical Benefit Rate (Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) > 4 Month)) - Per RECIST v1.1
Description: Phase II: Clinical Benefit Rate (Complete response (CR) or Partial response (PR) or Stable disease (SD) > 4 month)) per investigator based on Response evaluation criteria in solid tumors (RECIST) v1.1
Time Frame: 4 years
Population: Full Analysis Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 20 [7.1 to 40.1] | 0 [0.0 to 13.9] | 9.5 [1.7 to 27.1] | 10.0 [1.8 to 28.3]

5. Primary Outcome: Phase II: Bayesian Inference of Clinical Benefit Rate - Per RECIST v1.1- Mean
Description: as for outcome 4
Time Frame: 4 years
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per RECIST v1.1 - mean results | 0.8 [0 to 4.5] | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per RECIST v1.1 - mean results | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per RECIST v1.1 - mean results

6. Primary Outcome: Phase Ib: Planned Dose Intensity - MCS110
Description: To characterize the tolerability of MCS110 given in combination with PDR001 and to identify a recommended dose combination for Phase II. Planned dose intensity for MCS110 is cumulative planned dose (mg/kg)/ number of doses scheduled per protocol during treatment period (i.e., this is equivalent to planned dose level).
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Mean (Standard Deviation); unit: mg/kg/3wks
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
mg/kg/3wks | 0.86 (0.191) | 2.74 (0.386) | 2.66 (0.435) | 4.85 (0.286) | 7.05 (0.594) | 9.47 (1.093)

7. Primary Outcome: Phase Ib: Relative Dose Intensity - MCS110
Description: To characterize the tolerability of MCS110 given in combination with PDR001 and to identify a recommended dose combination for Phase II. Relative dose intensity (%) is 100 × dose intensity (mg/kg/3wks)/planned dose intensity (mg/kg/3wks).
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Percentage | 100 (100) | 100 (100) | 100 (100) | 99.23 (2.774) | 100 (100) | 100 (100)

8. Primary Outcome: Phase Ib: Planned Dose Intensity - PDR001
Description: To characterize the tolerability of MCS110 given in combination with PDR001 and to identify a recommended dose combination for Phase II. Planned dose intensity for PDR001 (mg/3wks) is planned cumulative dose (mg)/ number of doses scheduled per protocol during treatment period (i.e., this is equivalent to planned dose level).
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Mean (Standard Deviation); unit: mg/3wks
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
mg/3wks | 86.09 (19.058) | 91.18 (12.873) | 265.83 (43.528) | 293.59 (16.013) | 282.12 (23.773) | 289.04 (20.329)

9. Primary Outcome: Phase Ib: Relative Dose Intensity - PDR001
Description: To characterize the tolerability of MCS110 given in combination with PDR001 and to identify a recommended dose combination for Phase II. Relative dose intensity (%) is 100 × dose intensity (mg/3wks)/planned dose intensity (mg/3wks).
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Percentage | 100.00 (100.00) | 100.00 (100.00) | 100.00 (100.00) | 100.00 (100.00) | 100.00 (100.00) | 100.00 (100.00)

10. Primary Outcome: Phase Ib: Number of Participants With Dose Reductions
Description: To characterize the tolerability of MCS110 given in combination with PDR001 and to identify a recommended dose combination for Phase II.
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Participants
  n (%) of participants with no dose reduction- Study drug: MCS110 | 6 | 12 | 12 | 13 | 6 | 9
  n (%) of participants with no dose reduction- Study drug: PDR001 | 6 | 12 | 12 | 13 | 6 | 11

11. Primary Outcome: Phase Ib: Number of Dose Interruptions Per Participant
Description: as for outcome 10
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Mean (Standard Deviation); unit: Dose interruptions per participant
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Dose interruptions per participant
  Number of dose interruptions per subject - Study drug: MCS110 | 1.3 (1.97) | 0.3 (0.45) | 0.3 (0.45) | 0.0 (0.0) | 0.3 (0.52) | 0.1 (0.30)
  Number of dose interruptions per subject - Study drug: PDR001 | 1.3 (1.97) | 0.3 (0.45) | 0.3 (0.45) | 0.0 (0.0) | 0.3 (0.52) | 0.1 (0.30)

12. Primary Outcome: Phase Ib: Number of Subjects With at Least One Dose Interruption
Description: as for outcome 10
Time Frame: Measured up to a max of 112.4 weeks
Population: Safety Set. A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Participants
  Number of subjects with at least one dose interruption - by reason - Adverse Event - MCS110 | 3 | 3 | 3 | 0 | 2 | 1
  Number of subjects with at least one dose interruption - by reason - Adverse Event - PDR001 | 3 | 3 | 3 | 0 | 2 | 1

13. Primary Outcome: Phase Ib: Number of Participants With Dose Limiting Toxicities (DLTs) During the First 2 Cycles of Study Treatment
Description: Phase Ib: Dose limiting toxicities occurring during the first 2 cycles by system organ class, preferred term and maximum grade for Phase Ib. The National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 4.03 was used for all grading.
Time Frame: the first 2 cycles of study treatment; cycle = 21 days (i.e., at day 42)
Population: Dose Determination Set (DDS). A statistical analysis for this endpoint was not performed since it is not clinically relevant.
Measure: Count of Participants; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 5 | 11 | 9 | 7 | 4 | 4
Participants
  n (%) of subjects with at least one event - all grades | 0 | 0 | 1 | 0 | 0 | 1
  n (%) Investigations - all grades | 0 | 0 | 1 | 0 | 0 | 1
  n (%) Blood creatine phosphokinase increased - all grades | 0 | 0 | 1 | 0 | 0 | 1

14. Secondary Outcome: Phase II : Overall Response Rate (ORR) - Per irRC
Description: Phase II: Overall Response Rate (Complete response (CR) or Partial response (PR)) (with confirmation) as per investigator based on immune related Response criteria (irRC) (FAS)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 5 [0.3 to 21.6] | 0 [0.0 to 13.9] | 9.5 [1.7 to 27.1] | 0 [0.0 to 13.9]

15. Secondary Outcome: Phase Ib: Overall Response Rate (ORR)
Description: Phase Ib: Overall Response Rate (Complete response (CR) or Partial response (PR)), per RECIST v1.1 and per immune related Response criteria (irRC)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Percentage of participants
  Overall Response Rate as per investigator based on RECIST v1.1 | 16.7 [0.9 to 58.2] | 0 [0.0 to 22.1] | 0 [0.0 to 22.1] | 0 [0.0 to 20.6] | 0 [0.0 to 39.3] | 9.1 [0.5 to 36.4]
  Overall Response Rate - as per investigator based on irRC | 16.7 [0.9 to 58.2] | 0 [0.0 to 22.1] | 0 [0.0 to 22.1] | 0 [0.0 to 20.6] | 0 [0.0 to 39.3] | 9.1 [0.5 to 36.4]

16. Secondary Outcome: Phase II : Bayesian Inference of Overall Response Rate (ORR) - Per irRC - Mean
Description: Phase II: Overall Response Rate (Complete response (CR) or Partial response (PR)) (with confirmation) as per investigator based on immune related Response criteria (irRC)- mean (FAS)
Time Frame: 4 years
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 6.7 [0.8 to 17.1] | NA [NA to NA] — Bayesian inference of Clinical Benefit Rate was measured for this arm instead - see Bayesian inference of Clinical Benefit Rate - per irRC - mean results | 10.8 [2.6 to 23.1] | 0.8 [0 to 4.5]

17. Secondary Outcome: Phase 1b: Clinical Benefit Rate (CBR)
Description: Phase 1b: Clinical Benefit Rate (Complete response (CR) or Partial response (PR) or Stable disease (SD) > 4 month)) per RECIST v1.1 and per immune related Response criteria (irRC)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11
Percentage of participants
  Clinical Benefit Rate - as per investigator based on RECIST v1.1 | 33.3 [6.3 to 72.9] | 8.3 [0.4 to 33.9] | 0 [0.0 to 22.1] | 0 [0.0 to 20.6] | 0 [0.0 to 39.3] | 18.2 [3.3 to 47.0]
  Clinical Benefit Rate - as per investigator based on irRC | 50.0 [15.3 to 84.7] | 8.3 [0.4 to 33.9] | 0 [0.0 to 22.1] | 7.7 [0.4 to 31.6] | 33.3 [6.3 to 72.9] | 18.2 [3.3 to 47.0]

18. Secondary Outcome: Phase II: Clinical Benefit Rate (Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) > 4 Month)) - Per irRC
Description: Phase II: Clinical Benefit Rate (Complete response (CR) or Partial response (PR) or Stable disease (SD) > 4 month)) per immune related Response criteria (irRC)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | 20.0 [7.1 to 40.1] | 5.0 [0.3 to 21.6] | 19.0 [6.8 to 38.4] | 30.0 [14.0 to 50.8]

19. Secondary Outcome: Phase II: Bayesian Inference of Clinical Benefit Rate - Per irRC - Mean
Description: Phase II: Clinical Benefit Rate (Complete response (CR) or Partial response (PR) or Stable disease (SD) > 4 month)) per investigator based on immune related Response criteria (irRC)- mean (FAS)
Time Frame: 4 years
Population: as for outcome 3
Measure: Mean (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Percentage of participants | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per irRC - mean results | 5.6 [0.4 to 15.3] | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per irRC - mean results | NA [NA to NA] — Bayesian inference of Overall Response Rate was measured for this arm instead. See the Bayesian inference of Overall Response rate - per irRC - mean results

20. Secondary Outcome: Phase 1b and Phase II: Progression Free Survival Based on Investigator Assessment as Per RECIST v1.1 and Per Immune Related Response Criteria (irRC) - Using Kaplan-Meier Method - Median
Description: Phase 1b and Phase II: Progression Free Survival. Progression is defined as a 20% increase in the sum of diameter of measurable lesions taking as reference the smallest sum of diameter recorded at or after baseline, or worsening of non-measurable lesions or the appearance of new lesions, using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) or Per Immune Related Response Criteria (irRC). Unlike RECIST 1.1, PD per irRC requires confirmation at a new assessment after at least 4 weeks - using Kaplan-Meier method - Median.
Time Frame: Up to year 4
Population: Full Analysis Set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
months
  Median PFS - per RECIST v1.1 | 1.5 [1.1 to 14.8] | 1.3 [1.3 to 2.7] | 1.3 [0.8 to 1.3] | 1.1 [0.6 to 1.3] | 1.3 [0.5 to 4.0] | 1.2 [0.6 to 2.4] | 1.6 [1.4 to 2.8] | 1.3 [1.2 to 1.4] | 1.3 [1.2 to 1.4] | 2.4 [1.4 to 3.7]
  Median PFS - per iiRC | 8.2 [1.2 to 25.8] | 2.2 [1.3 to 2.7] | 1.3 [0.9 to 1.3] | 1.0 [0.5 to 1.3] | 1.3 [0.5 to 16.8] | 1.2 [0.7 to 2.4] | 1.6 [1.4 to 2.8] | 1.3 [1.2 to 1.5] | 1.3 [1.2 to 1.4] | 3.7 [1.4 to 4.2]

21. Secondary Outcome: Phase 1b and Phase II: Overall Survival - Using Kaplan-Meier Method - Median
Description: Phase 1b and Phase II: Overall Survival - using Kaplan-Meier method - Median
Time Frame: Up to year 4
Population: Full Analysis Set
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
months | 12.3 [3.1 to 26.6] | 9.6 [3.8 to 12.2] | 4.2 [1.5 to 7.9] | 2.8 [1.2 to 3.8] | 22.8 [1.1 to 26.8] | 5.7 [1.2 to 8.2] | 8.9 [5.6 to 16.6] | 2.6 [1.8 to 5.0] | 11.7 [9.2 to 14.6] | 19.7 [9.2 to 20.3]

22. Secondary Outcome: Phase 1b and Phase II: Duration of Response (DOR)
Description: Phase 1b and Phase II: Duration of Response (DOR) per RECIST v1.1 and per immune related Response criteria (irRC)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Median (Full Range); unit: days
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
days
  Duration of response(days) - based on RECIST v1.1 | 372.0 [372 to 372] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | 155.0 [155.0 to 155.0] | 169 [169 to 169] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | 328.5 [194 to 463] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median.
  Duration of response(days) - based on irRC | 372.0 [372.0 to 372.0] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | 155.0 [155.0 to 155.0] | 169 [169 to 169] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median. | 328.5 [194 to 463] | NA [NA to NA] — The median is not available because there was an insufficient number of participants with events. The lower and upper limits are not applicable since there is no value for median.

23. Secondary Outcome: Phase 1b and Phase II: Disease Control Rate (DCR)
Description: Phase 1b and Phase II: Disease Control Rate (Complete response (CR) or Partial response (PR) or Stable disease (SD) > 4 month)) per RECIST v1.1 and per immune related Response criteria (irRC)
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number (90% Confidence Interval); unit: Percentage
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Percentage
  Disease Control Rate - as per investigator based on RECIST v1.1 | 33.3 [6.3 to 72.9] | 8.3 [0.4 to 33.9] | 0 [0.0 to 22.1] | 15.4 [2.8 to 41.0] | 16.7 [0.9 to 58.2] | 18.2 [3.3 to 47.0] | 20.0 [7.1 to 40.1] | 0 [0.0 to 13.9] | 19.0 [6.8 to 38.4] | 35.0 [17.7 to 55.8]
  Disease Control Rate as per investigator based on irRC | 50.0 [15.3 to 84.7] | 8.3 [0.4 to 33.9] | 0 [0.0 to 22.1] | 15.4 [2.8 to 41.0] | 33.3 [6.3 to 72.9] | 18.2 [3.3 to 47.0] | 20.0 [7.1 to 40.1] | 5.0 [0.3 to 21.6] | 19.0 [6.8 to 38.4] | 45.0 [25.9 to 65.3]

24. Secondary Outcome: Phase II: Percentage of Participants With Adverse Events, as a Measure of Safety
Description: Phase II: To further characterize the safety and tolerability of MCS110 given in combination with PDR001
Time Frame: From start of treatment to a maximum timeframe of 92.4 weeks for phase II.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 20 | 20 | 21 | 20
Participants
  Adverse events - all grades | 20 | 20 | 21 | 20
  Adverse events - Treatment-related - all grades | 16 | 15 | 17 | 19
  SAEs - all grades | 8 | 14 | 8 | 7
  SAEs - Treatment-related - all grades | 1 | 4 | 4 | 1
  Fatal SAEs - all grades | 1 | 1 | 0 | 1
  Fatal SAEs - Treatment-related - all grades | 0 | 1 | 0 | 0
  AEs leading to discontinuation - all grades | 1 | 1 | 1 | 2
  AEs leading to discontinuation - Treatment-related - all grades | 1 | 0 | 1 | 1
  AEs leading to dose adjustment / interruption - all grades | 11 | 4 | 8 | 11
  AEs requiring additional therapy - all grades | 19 | 18 | 19 | 17

25. Secondary Outcome: Phase Ib and Phase II: Immunogenicity MCS110
Description: Phase Ib and Phase II: Presence of anti-MCS110 antibodies
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Participants
  Baseline positive | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative | 6 | 11 | 11 | 12 | 6 | 11 | 19 | 19 | 17 | 18
  Baseline missing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
  Baseline positive, on treatment persistent positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline positive, on treatment only last positive | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline positive, on treatment any positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline positive, on treatment all negative | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative, on treatment persistent positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative, on treatment only last positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative, on treatment any positive | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative, on treatment all negative | 5 | 10 | 8 | 6 | 5 | 6 | 12 | 16 | 14 | 17
  Baseline missing, on treatment persistent positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment only last positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment any positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment all negative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Phase Ib and Phase II: Immunogenicity PDR001
Description: Phase Ib and Phase II: Presence of anti-PDR001 antibodies
Time Frame: 4 years
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Participants
  Baseline positive | 0 | 2 | 1 | 2 | 1 | 2 | 1 | 1 | 0 | 1
  Baseline negative | 6 | 10 | 11 | 10 | 5 | 8 | 18 | 17 | 19 | 19
  Baseline missing | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 0
  Baseline positive, on treatment persistent positive | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline positive, on treatment only last positive | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Baseline positive, on treatment any positive | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
  Baseline positive, on treatment all negative | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline negative, on treatment persistent positive | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Baseline negative, on treatment only last positive | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 4 | 1 | 0
  Baseline negative, on treatment any positive | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Baseline negative, on treatment all negative | 4 | 4 | 8 | 6 | 4 | 2 | 11 | 10 | 16 | 13
  Baseline missing, on treatment persistent positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment only last positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment any positive | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Baseline missing, on treatment all negative | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1

27. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - AUClast and AUCinf
Description: Phase Ib and Phase II: PK Parameters - AUClast, which is the AUC from time zero to the last measurable concentration sampling time (tlast) (mass × time
  × volume-1); and AUCinf, which is the AUC from time zero to infinity (mass × time × volume-1) - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: Pharmacokinetic analysis set. Some patients were excluded because of missed visits, missed sampling, early termination, dosing outside the planned dose, or lost samples. There were some patients with AUClast but no AUCinf parameters because AUCinf could not be extrapolated from the data (i.e. the % of AUC extrapolated past the last time point is greater than 20% or the adjusted R squared parameter for the regression fit of the terminal phase of the PK profile is < 0.75).
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
day*ng/mL
  AUClast (day*ng/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 9 | 12 | 12 | 6 | 10 | 16 | 16 | 16 | 18
  AUClast (day*ng/mL) - cycle 1 - day 21 | 46900 (9080) | 343000 (142000) | 249000 (93400) | 490000 (149000) | 909000 (233000) | 1090000 (231000) | 1200000 (507000) | 1090000 (352000) | 1120000 (440000) | 1270000 (335000)
  AUCinf (day*ng/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 7 | 7 | 9 | 5 | 5 | 0 | 0 | 0 | 0
  AUCinf (day*ng/mL) - cycle 1 - day 21 | 50100 (11600) | 383000 (178000) | 330000 (73400) | 560000 (177000) | 1020000 (336000) | 988000 (116000) |  |  |  |
  AUClast (day*ng/mL) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 4 | 3 | 4 | 13
  AUClast (day*ng/mL) - cycle 4 - day 84 | 41000 (22800) | 213000 (92200) | 232000 (99300) | 710000 (171000) | 1520000 (353000) | 1200000 (1030000) | 1200000 (389000) | 918000 (102000) | 1010000 (337000) | 1240000 (499000)
  AUCinf (day*ng/mL) - cycle 4 - day 84: number analyzed (Participants) | 3 | 4 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  AUCinf (day*ng/mL) - cycle 4 - day 84 | 42300 (21900) | 260000 (73500) | 253000 (114000) | 619000 (NA) — SD is not applicable for an analysis with 1 participant |  | 769000 (NA) — SD is not applicable for an analysis with 1 participant |  |  |  |

28. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - AUClast and AUCinf
Description: Phase Ib and Phase II: Pharmacokinetics (PK) Parameters - AUClast, which is the AUC from time zero to the last measurable concentration sampling time (tlast) (mass × time
  × volume-1); and AUCinf, which is the AUC from time zero to infinity (mass × time × volume-1) and AUCinf - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 27
Measure: Mean (Standard Deviation); unit: day*ug/mL
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
day*ug/mL
  AUClast (day*ug/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 11 | 11 | 13 | 6 | 11 | 20 | 18 | 19 | 18
  AUClast (day*ug/mL) - cycle 1 - day 21 | 229 (68.3) | 271 (53.8) | 651 (322) | 604 (309) | 581 (147) | 450 (135) | 825 (402) | 782 (264) | 764 (311) | 782 (307)
  AUCinf (day*ug/mL) - cycle 1 - day 21: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  AUCinf (day*ug/mL) - cycle 1 - day 21 |  | 274 (NA) — SD is not applicable for an analysis with 1 participant | 610 (NA) — SD is not applicable for an analysis with 1 participant |  | 747 (NA) — SD is not applicable for an analysis with 1 participant | 710 (NA) — SD is not applicable for an analysis with 1 participant |  |  |  |
  AUClast (day*ug/mL) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 5 | 3 | 4 | 13
  AUClast (day*ug/mL) - cycle 4 - day 84 | 369 (26.4) | 330 (182) | 1020 (526) | 2020 (1170) | 954 (179) | 718 (288) | 1170 (388) | 1330 (555) | 1660 (283) | 1260 (533)
  AUCinf (day*ug/mL) - cycle 4 - day 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AUCinf (day*ug/mL) - cycle 4 - day 84 |  | 196 (NA) — SD is not applicable for an analysis with 1 participant |  |  |  |  |  |  |  |

29. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - Cmax and Clast
Description: Phase Ib and Phase II: PK Parameters - Cmax, which is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass × volume-1); and Clast - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: Pharmacokinetic analysis set. Some patients were excluded from the PK parameter analysis because of missed visits, missed sampling, early termination, dosing outside the planned dose, or lost samples.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
ng/mL
  Cmax (ng/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 9 | 12 | 12 | 6 | 10 | 16 | 16 | 16 | 18
  Cmax (ng/mL) - cycle 1 - day 21 | 17400 (1870) | 58800 (16900) | 56700 (17800) | 96900 (28600) | 122000 (17100) | 186000 (54000) | 158000 (44800) | 130000 (38400) | 134000 (64900) | 151000 (42500)
  Clast (ng/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 9 | 12 | 12 | 6 | 10 | 16 | 16 | 16 | 18
  Clast (ng/mL) - cycle 1 - day 21 | 1120 (795) | 1290 (2760) | 6600 (6370) | 9130 (11500) | 15100 (9070) | 28700 (27800) | 33000 (21300) | 12900 (10700) | 24500 (20100) | 17500 (11400)
  Cmax (ng/mL) -- cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 4 | 3 | 4 | 13
  Cmax (ng/mL) -- cycle 4 - day 84 | 13500 (5580) | 53000 (9790) | 48900 (14100) | 76400 (24000) | 176000 (19800) | 189000 (29400) | 159000 (39800) | 152000 (58000) | 128000 (42600) | 147000 (38300)
  Clast (ng/mL) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 4 | 3 | 4 | 13
  Clast (ng/mL) - cycle 4 - day 84 | 510 (457) | 5700 (10300) | 3490 (2410) | 7350 (5870) | 45100 (12400) | 34100 (29800) | 57600 (45000) | 33300 (42600) | 18600 (21700) | 29400 (20700)

30. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - Cmax and Clast
Description: Phase Ib and Phase II: PK Parameters - Cmax, which is the maximum (peak) observed plasma, blood, serum, or other body fluid drug concentration after single dose administration (mass × volume-1); and Clast - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
ug/mL
  Cmax (ug/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 11 | 11 | 13 | 6 | 11 | 20 | 18 | 19 | 18
  Cmax (ug/mL) - cycle 1 - day 21 | 24 (9.52) | 29.5 (6.56) | 73.4 (22.3) | 77 (24.3) | 76.6 (36.8) | 64.2 (20.4) | 94.5 (27.4) | 75.3 (23.9) | 80.2 (24) | 70.3 (21.6)
  Clast (ug/mL) - cycle 1 - day 21: number analyzed (Participants) | 6 | 11 | 11 | 13 | 6 | 11 | 20 | 18 | 19 | 18
  Clast (ug/mL) - cycle 1 - day 21 | 7.73 (2.97) | 7.24 (2.95) | 19.4 (11.7) | 26.4 (11.8) | 22.7 (12.8) | 17.2 (8.67) | 34.5 (13.3) | 24 (12) | 22.8 (9.44) | 24.4 (14.6)
  Cmax (ug/mL) -- cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 5 | 3 | 4 | 13
  Cmax (ug/mL) -- cycle 4 - day 84 | 29.5 (9.3) | 36.8 (10.5) | 126 (54.6) | 153 (22.6) | 92 (22.1) | 85.9 (16.8) | 123 (56.8) | 127 (7) | 122 (23.6) | 108 (23.4)
  Clast (ug/mL) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 5 | 3 | 4 | 13
  Clast (ug/mL) - cycle 4 - day 84 | 10.7 (2.25) | 14.5 (8.47) | 65.1 (37.6) | 71 (6.65) | 47.5 (25.7) | 35.6 (14.7) | 81.4 (43.6) | 62.1 (9.93) | 48.8 (20.6) | 51.3 (23.7)

31. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - Tmax
Description: Phase Ib and Phase II: PK Parameters - Tmax, which is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time) - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Median (Full Range); unit: hour
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
hour
  Tmax (h) - cycle 1 - day 21: number analyzed (Participants) | 6 | 9 | 12 | 12 | 6 | 10 | 16 | 16 | 16 | 18
  Tmax (h) - cycle 1 - day 21 | 2.02 [1.5 to 2.08] | 1.92 [0.5 to 23.7] | 2.08 [1.5 to 22.2] | 2.13 [1.92 to 24] | 2.06 [2 to 24.4] | 2.04 [1.92 to 26.2] | 2.01 [0.5 to 162] | 2.08 [1.92 to 2.28] | 2.09 [2 to 163] | 2.08 [1.5 to 188]
  Tmax (h) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 4 | 3 | 4 | 13
  Tmax (h) - cycle 4 - day 84 | 2 [2 to 2] | 2.05 [0.5 to 2.08] | 2.03 [2 to 23.7] | 13 [2.02 to 24] | 2 [2 to 20.8] | 2.03 [1.98 to 21.3] | 2 [1.92 to 2.12] | 2.02 [1.98 to 2.08] | 2.04 [2 to 2.12] | 2.05 [2 to 2.13]

32. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - Tmax
Description: Phase Ib and Phase II: PK Parameters - Tmax, which is the time to reach maximum (peak) plasma, blood, serum, or other body fluid drug concentration after single dose administration (time) - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Median (Full Range); unit: hour
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
hour
  Tmax (h) - cycle 1 - day 21: number analyzed (Participants) | 6 | 11 | 11 | 13 | 6 | 11 | 20 | 18 | 19 | 18
  Tmax (h) - cycle 1 - day 21 | 11.5 [1.48 to 26] | 2.08 [1.5 to 25.5] | 1.53 [1 to 26.5] | 1.57 [1.5 to 22.3] | 1.53 [0.983 to 25.8] | 1.52 [1.5 to 22.8] | 1.5 [1 to 168] | 1.5 [0.5 to 3.22] | 1.5 [1.42 to 166] | 1.5 [1.45 to 624]
  Tmax (h) - cycle 4 - day 84: number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 5 | 3 | 4 | 13
  Tmax (h) - cycle 4 - day 84 | 1.52 [1.5 to 22.4] | 1.53 [0 to 23.7] | 1.2 [0 to 1.5] | 1.57 [1.55 to 1.58] | 1.5 [1.5 to 3.42] | 1.45 [1.43 to 2.92] | 1.53 [1.5 to 165] | 1.47 [1.42 to 1.48] | 1.54 [1.48 to 1.62] | 1.5 [1.43 to 1.67]

33. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - T1/2
Description: Phase Ib and Phase II: PK Parameters - T1/2, which is the terminal half-life associated with the terminal slope of a semi logarithmic concentration time curve (time) - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Median (Full Range); unit: day
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
day
  T1/2 (day) - cycle 1 - day 21: number analyzed (Participants) | 6 | 7 | 7 | 9 | 5 | 5 | 0 | 0 | 0 | 0
  T1/2 (day) - cycle 1 - day 21 | 1.5 [1.25 to 2.38] | 2.16 [1.68 to 6.71] | 3.3 [1.85 to 5.32] | 3.48 [1.73 to 7.82] | 6.35 [2.17 to 8.05] | 4.36 [2.25 to 6.62] |  |  |  |
  T1/2 (day) - cycle 4 - day 84: number analyzed (Participants) | 3 | 4 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  T1/2 (day) - cycle 4 - day 84 | 1.77 [1.23 to 1.81] | 1.53 [1.03 to 2.49] | 4.08 [1.41 to 4.26] | 6.32 [6.32 to 6.32] |  | 4.82 [4.82 to 4.82] |  |  |  |

34. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - T1/2
Description: Phase Ib and Phase II: PK Parameters - T1/2, which is the terminal half-life associated with the terminal slope of a semi logarithmic concentration time curve (time) - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Median (Full Range); unit: day
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
day
  T1/2 (day) - cycle 1 - day 21: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  T1/2 (day) - cycle 1 - day 21 |  | 8.14 [8.14 to 8.14] | 7.71 [7.71 to 7.71] |  | 7.13 [7.13 to 7.13] | 7.33 [7.33 to 7.33] |  |  |  |
  T1/2 (day) - cycle 4 - day 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  T1/2 (day) - cycle 4 - day 84 |  | 7.81 [7.81 to 7.81] |  |  |  |  |  |  |  |

35. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - CL
Description: Phase Ib and Phase II: PK Parameters - CL, which is the total body clearance of drug from the plasma (volume × time-1) - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: L/h/kg
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
L/h/kg
  CL (L/h/kg) - cycle 1 - day 21: number analyzed (Participants) | 6 | 7 | 7 | 9 | 5 | 5 | 0 | 0 | 0 | 0
  CL (L/h/kg) - cycle 1 - day 21 | 0.000863 (0.000158) | 0.000388 (0.000181) | 0.000394 (0.0000833) | 0.000407 (0.000131) | 0.000338 (0.000117) | 0.000427 (0.0000558) |  |  |  |
  CL (L/h/kg) - cycle 4 - day 84: number analyzed (Participants) | 3 | 4 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  CL (L/h/kg) - cycle 4 - day 84 | 0.00117 (0.000549) | 0.000523 (0.000199) | 0.000315 (0.000218) | 0.000337 (NA) — Not Evaluable |  | 0.000541 (NA) — Not Evaluable |  |  |  |

36. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - CL
Description: Phase Ib and Phase II: PK Parameters - CL, which is the total body clearance of drug from the plasma (volume × time-1) - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
L/h
  CL (L/h) - cycle 1 - day 21: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  CL (L/h) - cycle 1 - day 21 |  | 0.0152 (NA) — Not Evaluable | 0.0205 (NA) — Not Evaluable |  | 0.0167 (NA) — Not Evaluable | 0.0176 (NA) — Not Evaluable |  |  |  |
  CL (L/h) - cycle 4 - day 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CL (L/h) - cycle 4 - day 84 |  | 0.0213 (NA) — Not Evaluable |  |  |  |  |  |  |  |

37. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - Vz
Description: Phase Ib and Phase II: PK Parameters - Vz, which is the apparent volume of distribution during terminal phase (volume) - MCS110
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: L/kg
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
L/kg
  Vz (L/kg) - cycle 1 - day 21: number analyzed (Participants) | 6 | 7 | 7 | 9 | 5 | 5 | 0 | 0 | 0 | 0
  Vz (L/kg) - cycle 1 - day 21 | 0.0486 (0.00989) | 0.0334 (0.00783) | 0.0423 (0.00875) | 0.051 (0.0206) | 0.0651 (0.0201) | 0.065 (0.0267) |  |  |  |
  Vz (L/kg) - cycle 4 - day 84: number analyzed (Participants) | 3 | 4 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Vz (L/kg) - cycle 4 - day 84 | 0.0684 (0.0407) | 0.0294 (0.0128) | 0.045 (0.0308) | 0.0736 (NA) — Not Evaluable |  | 0.0904 (NA) — Not Evaluable |  |  |  |

38. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - Vz
Description: Phase Ib and Phase II: PK Parameters - Vz, which is the apparent volume of distribution during terminal phase (volume) - PDR001
Time Frame: cycle 1 (day 21) and cycle 4 (day 84)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Liters (L)
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 11 | 12 | 13 | 6 | 11 | 20 | 19 | 20 | 20
Liters (L)
  Vz (L) - cycle 1 - day 21: number analyzed (Participants) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
  Vz (L) - cycle 1 - day 21 |  | 4.28 (NA) — Not Evaluable | 5.47 (NA) — Not Evaluable |  | 4.13 (NA) — Not Evaluable | 4.47 (NA) — Not Evaluable |  |  |  |
  Vz (L) - cycle 4 - day 84: number analyzed (Participants) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Vz (L) - cycle 4 - day 84 |  | 5.76 (NA) — Not Evaluable |  |  |  |  |  |  |  |

39. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of MCS110 - Accumulation Ratio (AR)
Description: Phase Ib and Phase II: PK Parameters - Accumulation ratio (AR), which is the AUClast (multiple Dose)/AUClast (single dose) (for cycle 4 only) - MCS110
Time Frame: cycle 4 (day 84)
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: Ratio of AUC
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 4 | 3 | 4 | 12
Ratio of AUC | 0.789 (0.232) | 0.744 (0.307) | 0.833 (0.0739) | 1.14 (0.0991) | 1.37 (0.278) | 1.04 (0.731) | 0.712 (0.205) | 0.829 (0.177) | 0.723 (0.315) | 0.987 (0.35)

40. Secondary Outcome: Phase Ib and Phase II: Pharmacokinetics of PDR001 - Accumulation Ratio (AR)
Description: Phase Ib and Phase II: PK Parameters - Accumulation ratio (AR), which is the AUClast (multiple Dose)/AUClast (single dose) (for cycle 4 only) - PDR001
Time Frame: cycle 4 (day 84)
Population: Pharmacokinetic analysis set
Measure: Mean (Standard Deviation); unit: Ratio of AUC
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 3 | 6 | 4 | 2 | 3 | 3 | 5 | 3 | 4 | 13
Ratio of AUC | 1.48 (0.17) | 1.15 (0.522) | 1.14 (0.176) | 1.89 (0.84) | 1.85 (0.348) | 1.5 (0.848) | 1.08 (0.235) | 1.56 (0.593) | 2.05 (0.156) | 1.54 (0.664)

41. Secondary Outcome: Phase Ib and Phase II: All Collected Deaths
Description: On treatment deaths are reported from the start of treatment until end of study treatment plus 30 days, up to maximum duration of 116.4 weeks for phase Ib and 92.4 weeks for phase II. Deaths post treatment survival follow up are reported after the on-treatment period, up to a maximum timeframe of 46 months (3.8 years).
Time Frame: For ontreatment deaths: up to maximum timeframe of 116.4 weeks for phase Ib and 92.4 weeks for phase II. For total deaths: up to 3.8 years
Population: Clinical Database Population
Measure: Number; unit: Participants
Arm/Group | Ph Ib: MCS110 1 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 100 mg Q3W | Ph Ib: MCS110 3 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W | Ph Ib: MCS110 10 mg/kg Q3W + PDR001 300 mg Q3W | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - TNBC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - PC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - EC | Ph II: MCS110 7.5 mg/kg Q3W + PDR001 300 mg Q3W - ME
Number analyzed (Participants) | 6 | 12 | 12 | 13 | 6 | 11 | 20 | 20 | 21 | 20
Participants
  Total Deaths | 6 | 12 | 10 | 12 | 4 | 10 | 11 | 19 | 14 | 11
  On-treatment Deaths | 0 | 1 | 4 | 4 | 1 | 4 | 1 | 3 | 0 | 2

ADVERSE EVENTS:
Time Frame: On-treatment adverse events are reported, from first dose of study treatment until end of study treatment plus 30 days, up to maximum timeframe of 116.4 weeks for phase Ib and 92.4 weeks for phase II.
Groups:
- Ph Ib: MCS110@1 mg/kg Q3W@+ PDR001 100@mg Q3W: Ph Ib: MCS110@1 mg/kg Q3W@+ PDR001 100@mg Q3W
- Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 100@mg Q3W: Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 100@mg Q3W
- Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 300@mg Q3W: Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 300@mg Q3W
- Ph Ib: MCS110@5 mg/kg Q3W@+ PDR001 300@mg Q3W: Ph Ib: MCS110@5 mg/kg Q3W@+ PDR001 300@mg Q3W
- Ph Ib: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W: Ph Ib: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W
- Ph Ib: MCS110@10 mg/kg Q3W@+ PDR001 300@mg Q3W: Ph Ib: MCS110@10 mg/kg Q3W@+ PDR001 300@mg Q3W
- Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - TNBC: Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - TNBC
- Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - PC: Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - PC
- Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - EC: Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - EC
- Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - ME: Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - ME
Arm/Group | Ph Ib: MCS110@1 mg/kg Q3W@+ PDR001 100@mg Q3W | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 100@mg Q3W | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 300@mg Q3W | Ph Ib: MCS110@5 mg/kg Q3W@+ PDR001 300@mg Q3W | Ph Ib: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W | Ph Ib: MCS110@10 mg/kg Q3W@+ PDR001 300@mg Q3W | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - TNBC | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - PC | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - EC | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - ME
All-Cause Mortality (participants affected / at risk) | 0/6 | 1/12 | 4/12 | 4/13 | 1/6 | 4/11 | 1/20 | 3/20 | 0/21 | 2/20
Serious Adverse Events (participants affected / at risk) | 3/6 | 4/12 | 4/12 | 7/13 | 2/6 | 5/11 | 8/20 | 14/20 | 8/21 | 7/20
Other Adverse Events (participants affected / at risk) | 6/6 | 12/12 | 12/12 | 13/13 | 6/6 | 11/11 | 20/20 | 20/20 | 21/21 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ph Ib: MCS110@1 mg/kg Q3W@+ PDR001 100@mg Q3W (N=6) | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 100@mg Q3W (N=12) | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 300@mg Q3W (N=12) | Ph Ib: MCS110@5 mg/kg Q3W@+ PDR001 300@mg Q3W (N=13) | Ph Ib: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W (N=6) | Ph Ib: MCS110@10 mg/kg Q3W@+ PDR001 300@mg Q3W (N=11) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - TNBC (N=20) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - PC (N=20) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - EC (N=21) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - ME (N=20)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device breakage (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ph Ib: MCS110@1 mg/kg Q3W@+ PDR001 100@mg Q3W (N=6) | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 100@mg Q3W (N=12) | Ph Ib: MCS110@3 mg/kg Q3W@+ PDR001 300@mg Q3W (N=12) | Ph Ib: MCS110@5 mg/kg Q3W@+ PDR001 300@mg Q3W (N=13) | Ph Ib: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W (N=6) | Ph Ib: MCS110@10 mg/kg Q3W@+ PDR001 300@mg Q3W (N=11) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - TNBC (N=20) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - PC (N=20) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - EC (N=21) | Ph II: MCS110@7.5 mg/kg Q3W@+ PDR001 300@mg Q3W - ME (N=20)
Anaemia (Blood and lymphatic system disorders) | 4 | 2 | 3 | 3 | 3 | 3 | 4 | 6 | 5 | 7
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 3 | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 4 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Panophthalmitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 3 | 2 | 1 | 1 | 0 | 3 | 3 | 4 | 6
Uveitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Xerophthalmia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 3 | 3 | 1 | 1 | 0 | 3 | 3 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 2 | 2 | 2 | 1 | 6 | 4 | 4 | 5
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 0 | 1 | 2 | 3 | 2 | 4 | 2 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 5 | 3 | 5 | 1 | 6 | 6 | 8 | 6 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5 | 3 | 5 | 1 | 1 | 3 | 4 | 2 | 0
Adverse reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 3 | 5 | 3 | 3 | 3 | 5 | 2 | 3 | 2 | 3
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 4 | 3 | 7
Face oedema (General disorders) | 0 | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 3 | 6
Fatigue (General disorders) | 2 | 3 | 5 | 2 | 2 | 0 | 5 | 2 | 4 | 4
Gait disturbance (General disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Generalised oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 3 | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1
Oedema peripheral (General disorders) | 2 | 1 | 2 | 2 | 1 | 1 | 2 | 3 | 3 | 3
Pyrexia (General disorders) | 1 | 4 | 3 | 1 | 0 | 5 | 4 | 4 | 1 | 8
Suprapubic pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Helicobacter infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Otitis media (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Pyuria (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 0
Viral skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 0 | 1 | 1 | 3 | 2 | 3 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post procedural inflammation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 2 | 1 | 1 | 2 | 4 | 5 | 7 | 4
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 3 | 5 | 3 | 4 | 9 | 7 | 13 | 10
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 3 | 2 | 0 | 0 | 2 | 3 | 3 | 3
Blood bilirubin increased (Investigations) | 3 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3 | 3 | 3 | 4 | 3 | 9 | 10 | 12 | 14
Blood creatinine increased (Investigations) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 5
Blood pressure increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 1
Neutrophil count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 7 | 4 | 1 | 0 | 4 | 3 | 7 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 1 | 1 | 0 | 0 | 3 | 2 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 4 | 2 | 1 | 0 | 1 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint warmth (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 4 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 5 | 0 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 3 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eating disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 1
Choluria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 1 | 0 | 2 | 1 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal mucosal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 1 | 0 | 2 | 2 | 2 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 0 | 1 | 1 | 3 | 2 | 2 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT02807844/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/44/NCT02807844/SAP_001.pdf